CLINICAL TRIAL: NCT04656288
Title: A Two-part Phase I Trial Investigating the Relative Bioavailability and Food Effect of Different Oral Formulations of BI 764198 in Healthy Subjects (an Open-label, Single-dose, Randomised, Crossover Study)
Brief Title: A Study in Healthy Men to Test if Different Formulations of BI 764198 With or Without Food Influence the Amount of BI 764198 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1434-0010; 2020-004757-79 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Formula A under fasted conditions - Part 1 (Experimental)
  Interventions: Drug: BI 764198 - Formula A
- Formula B under fasted conditions - Part 1 (Experimental)
  Interventions: Drug: BI 764198 - Formula B
- Formula B under fasted conditions - Part 2 (Experimental)
  Interventions: Drug: BI 764198 - Formula B
- Formula C under fasted conditions - Part 2 (Experimental)
  Interventions: Drug: BI 764198 - Formula C
- Formula D under fasted conditions - Part 2 (Experimental)
  Interventions: Drug: BI 764198 - Formula D
- Formula B under fed conditions - Part 2 (Experimental)
  Interventions: Drug: BI 764198 - Formula B

INTERVENTIONS:
Drug: BI 764198 - Formula A — BI 764198
  Arms: Formula A under fasted conditions - Part 1
Drug: BI 764198 - Formula B — BI 764198
  Arms: Formula B under fasted conditions - Part 1; Formula B under fasted conditions - Part 2; Formula B under fed conditions - Part 2
Drug: BI 764198 - Formula C — BI 764198
  Arms: Formula C under fasted conditions - Part 2
Drug: BI 764198 - Formula D — BI 764198
  Arms: Formula D under fasted conditions - Part 2

SUMMARY:
BI 764198 is intended to be used in patients hospitalized for COVID-19 at risk of respiratory complications. The present trial will investigate the relative bioavailability of BI 764198 administered as capsules versus tablets in a first part, and the relative bioavailability and food effect of four oral formulations: the newly developed tablet formulation under fed and fasted conditions as well as suspension from capsules and suspension from tablets in a second part.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive) at screening
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive) at screening
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who meet any of the following criteria from first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception by the female partners, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device that started at least 2 months prior to first drug administration to the male subject, or barrier method (e.g. diaphragm with spermicide), or surgically sterilised (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy), or postmenopausal, defined as at least 1 year of spontaneous amenorrhea
  * Sexually abstinent
  * Vasectomised (vasectomy at least 1 year prior to enrolment) in combination with a barrier method (e.g. condom) Sperm donation is not allowed from first study drug administration until 30 days after trial completion.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Part 1: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 4 days per period
Part 1: Cmax (maximum measured concentration of the analyte in plasma) | up to 4 days per period
Part 2: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 5 days per period
Part 2: Cmax (maximum measured concentration of the analyte in plasma) | up to 5 days per period

SECONDARY OUTCOMES:
Part 1: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 4 days per period
Part 2: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 5 days per period

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Belgium NV Research Unit Stuivenberg, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Schultz A, Halabi A, Seitz F, Lemmens K, Wulfrath HS, Lobmeyer MT, Retlich S, Choi W, Soleymanlou N. Phase 1 trials of BI 764198, a transient receptor potential channel 6 inhibitor, in healthy volunteers and participants with kidney impairment. Expert Opin Investig Drugs. 2025 May;34(5):415-423. doi: 10.1080/13543784.2025.2510673. Epub 2025 Jun 8. PMID 40455255
- See also: Related Info — https://www.mystudywindow.com/